CLINICAL TRIAL: NCT05348980
Title: Comparison of Two Different Doses of Intramuscular Phenylephrine HCL for Prevention of Spinal Anesthesia Induced Hypotension During Cesarean Section: A Prospective Randomized Double-blinded Parallel Study
Brief Title: Intramuscular Phenylephrine HCL for Prevention of Spinal Anesthesia Induced Hypotension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rehman Medical Institute - RMI (Other)
Responsible Party: Principal Investigator, Mohammad Shafiq, Principal investigator, Rehman Medical Institute - RMI
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RMI/RMI-REC/Approval/57
Record Dates: First submitted 2022-04-04; First posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Hypotension; Anesthesia
Keywords: Cesarean section.
MeSH Terms: conditions — Hypotension | interventions — Phenylephrine

STUDY DESIGN:
Intervention Model Description: The study design was prospective double-blinded randomized parallel with allocation ratio of 1:1.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Two color coded envelops containing drug doses for intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phenylephrine 4mg (Active Comparator): Inj Phenylephrine HCL 04 mg as Group P4.
  Interventions: Drug: Phenylephrine Hydrochloride 4 mg
- Phenylephrine 8mg (Active Comparator): Inj Phenylephrine HCL 08 mg as Group P8.
  Interventions: Drug: Phenylephrine Hydrochloride 8 mg

INTERVENTIONS:
Drug: Phenylephrine Hydrochloride 4 mg — Intramuscular Phenylephrine HCL 04 mg were administered as prophylactic stat dose in Vastus lateralis muscle of thigh 05 minutes before giving spinal anesthesia.
  Other Names: Injection Synephrine (Atco Laboratories Ltd. Pakistan
  Arms: Phenylephrine 4mg
Drug: Phenylephrine Hydrochloride 8 mg — Intramuscular Phenylephrine HCL 08 mg were administered as prophylactic stat dose in Vastus lateralis muscle of thigh 05 minutes before giving spinal anesthesia.
  Other Names: Injection Synephrine (Atco Laboratories Ltd. Pakistan
  Arms: Phenylephrine 8mg

SUMMARY:
Background: Spinal anesthesia (SA) is preferred over general anesthesia in Cesarean section (CS) due to its better safety profile but SA induced hypotension remains a big challenge for the clinical Anesthetist. Different methods including 15° left lateral table tilt, leftward uterine manual displacement, fluid pre-and co-loading have been used but drop in Systolic Blood Pressure (SBP) jeopardizing maternal and fetal well-being still occurs. Timely administered Phenylephrine HCL, an α-1 adrenergic agonist, is a recommended remedy.

Subjects and methods: Sixty parturients of American Society of Anaesthesiologists (ASA) physical status 1 and 2, scheduled for elective CS under SA were enrolled in this prospective double-blinded study and randomly divided into two equal groups, P4 and P8. They received intramuscular (IM) Phenylephrine HCL 04 mg and 08 mg respectively before SA. Spinal block up to T6 was achieved with 12.5 mg 0.5% Bupivacaine HCl heavy. The incidence and intensity of hypotension, rescue doses of Phenylephrine HCL and any adverse event, were recorded. Data collected was analyzed using Epi lnfo ™ version 7.2.

DETAILED DESCRIPTION:
Introduction: World Health Organization (WHO) defines maternal death as a death while pregnant or within 42 days of the end of gestation, from any cause related to or aggravated by the pregnancy or its management (excluding accidental or incidental causes). In 2017 global Maternal Mortality Ratio (MMR) reported by United Nations (UN) is 211 deaths per 100,000 live births. MMR in Pakistan, with inter-provincial variability, is 186 deaths per 100,000 live births according to the latest Pakistan Maternal Mortality Survey (PMMS) report published in August, 2020 by United Nations Population Fund (UNFPA), a subsidiary organ of United Nations General Assembly.

CS requires general anesthesia, SA or epidural anesthesia; however, SA is preferred. SA is believed to be safe, though severe complications like profound hypotension compounded by aorto-caval compression might happen . World Health Organization (WHO) defines ideal CS rate below 10 to 15 %. According to 1990-91 and 2017-18 Pakistan Demographic and Health Survey data, rate of C-section has been raised from 3.2 % to 19.6 - 22.3 % . Higher rate of anesthesia and surgery in a developing country like Pakistan has a direct bearing on MMR, patient's morbidity, cost of medical services and siphoning scarce resources.

The first case of cardiac arrest occurring after SA was reported in 1940 and since then, the ability of SA to cause cardio-pulmonary arrest was considered. Hypotension and bradycardia are the most common side effects of SA. SA induced hypotension, which is a substantial clinical challenge, is caused by pharmacological sympathectomy. The incidence is reported around 80 %. Hypotension occurs despite fluid preload, left lateral uterine displacement and left lateral table tilt.

Duration and severity of hypotension is responsible for maternal ill effects like nausea/vomiting initially and later culminating to dyspnoea, apnea and circulatory arrest if poorly managed. Additionally there will be poor apgar score or even fetal demise depending upon the severity. Energetic use of strong vasopressors has been recommended. Phenylephrine HCL is considered to be the vasopressor of choice in parturients due to its propensity to cause less fetal acidosis. Phenylephrine HCL being an α-1adrenergic agonist counters the decrease in Systemic Vascular Resistance (SVR) induced by SA and can be administered by subcutaneous, intravenous and IM routes. Its onset and duration of action are 1-3 minutes and 5- 20 minutes respectively, when given intravenously (IV); and 10-20 minutes and an hour respectively when given IM. Clinically, 50-100 microgram boluses of Phenylephrine HCL is used intravenously to address hypotension. The investigators, in the current study exploited its lesser reported IM route.

Rationale: IM Phenylephrine HCL shortly before administering SA can prove a better option to prevent hypotension even for longer duration due to its slower absorption and can provide longer hemodynamic stability, lesser drop in fetal pH and apgar score.

Objectives: The primary objective of the study was to determine appropriate dose of IM Phenylephrine HCL in preventing hypotension due to SA administered for CS in ASA 1 and 2 parturients. Secondary objectives were to determine the need for total rescue doses of Phenylephrine HCL, measure drop in SBP in the two trial groups; and observe any side effects associated with IM injection of Phenylephrine HCL.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant ladies of American Society of Anesthesiologists (ASA) physical status 1 or 2 with
* Singleton Pregnancy,
* Full term pregnancy, and
* Admitted for elective CS

Exclusion Criteria:

All those participants having;

* Blood pressure ≥140/90 mm of Hg,
* ASA 3 or above status,
* Contraindication to spinal anesthesia
* Fetal anomalies/
* Abnormal placentae
* Refusal to consent

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Incidence of hypotension in both groups | One and half hour post spinal anesthesia
  The primary outcome is to find incidence of hypotension in each group P4 and P8 i.e. number of participants who develop hypotension in the relevant group multiplied by 100.
  Incidence= number of participants who develop hypotension/ total participants in the group *100.
  Hypotension is defined as a decrease of more than 20 % from baseline systolic blood pressure measured through non-invasive method.

SECONDARY OUTCOMES:
To find the rescue dose/ doses of intravenous Phenylephrine HCL. | One and half hour post spinal anesthesia
  To find the rescue dose/ doses of intravenous Phenylephrine in the two groups P4 and P8.
Onset of hypotension | Half hour/ 30 minutes post spinal anesthesia
  Determine the onset of hypotension in the two groups P4 and P8 (keeping starting time 0 minute at the administration of intrathecal hyperbaric Bupivacaine).
Adverse events associated with any groups | One and half hour post spinal anesthesia
  Record any adverse event associated with any groups e.g. bradycardia, hypotension, Nausea, Vomiting, Hypertension, Cardiac arrest.
Neonatal APGAR Score | 5 minutes post delivery
  Neonatal APGAR (Appearance, Pulse, Grimace response, Activity, and Respiration)Score from 0 - 10 will be measured at 01 and 05 minutes for each neonate delivered. The higher score is considered good i.e. 10 while lower score is considered bad/ worse e.g. 0 -3.
  The Apgar score measures five things to check a baby's health. Each is scored on a scale of 0 to 2, with 2 being the best score:
  Appearance (skin color) Pulse (heart rate) Grimace response (reflexes) Activity (muscle tone) Respiration (breathing rate and effort)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Shafiq, FCPS, Principal Investigator — Rehman Medical Institute
Locations (1):
- Rehman Medical Institute, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Data including clinical and demographic characteristics, not affecting patient's confidentiality, will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: April, 2022 to April, 2025.
Access Criteria: IPD will be shared on inter institutional request basis.

REFERENCES:
- [Background] Shitemaw T, Jemal B, Mamo T, Akalu L. Incidence and associated factors for hypotension after spinal anesthesia during cesarean section at Gandhi Memorial Hospital Addis Ababa, Ethiopia. PLoS One. 2020 Aug 13;15(8):e0236755. doi: 10.1371/journal.pone.0236755. eCollection 2020. PMID 32790681
- [Background] Michelsen TM, Tronstad C, Rosseland LA. Blood pressure and cardiac output during caesarean delivery under spinal anaesthesia: a prospective cohort study. BMJ Open. 2021 Jun 14;11(6):e046102. doi: 10.1136/bmjopen-2020-046102. PMID 34127491
- [Background] Richards E, Lopez MJ, Maani C V. Phenylephrine. xPharm Compr Pharmacol Ref [Internet]. 2021 Jul 13 [cited 2022 Jan 17];1-5. Available from: https://www.ncbi.nlm.nih.gov/books/NBK534801/
- [Result] GBD 2015 Maternal Mortality Collaborators. Global, regional, and national levels of maternal mortality, 1990-2015: a systematic analysis for the Global Burden of Disease Study 2015. Lancet. 2016 Oct 8;388(10053):1775-1812. doi: 10.1016/S0140-6736(16)31470-2. PMID 27733286
- [Result] Amjad A, Imran A, Shahram N, Zakar R, Usman A, Zakar MZ, Fischer F. Trends of caesarean section deliveries in Pakistan: secondary data analysis from Demographic and Health Surveys, 1990-2018. BMC Pregnancy Childbirth. 2020 Dec 2;20(1):753. doi: 10.1186/s12884-020-03457-y. PMID 33267787
- [Result] Ferre F, Martin C, Bosch L, Kurrek M, Lairez O, Minville V. Control of Spinal Anesthesia-Induced Hypotension in Adults. Local Reg Anesth. 2020 Jun 3;13:39-46. doi: 10.2147/LRA.S240753. eCollection 2020. PMID 32581577
- [Result] Rijs K, Mercier FJ, Lucas DN, Rossaint R, Klimek M, Heesen M. Fluid loading therapy to prevent spinal hypotension in women undergoing elective caesarean section: Network meta-analysis, trial sequential analysis and meta-regression. Eur J Anaesthesiol. 2020 Dec;37(12):1126-1142. doi: 10.1097/EJA.0000000000001371. PMID 33109924
- [Result] EVALUATION OF PREEMPTIVE INTRAMUSCULAR EPHEDRINE VS PHENYLEPHRINE IN PREVENTION OF HYPOTENSION INDUCED BY SPINAL ANESTHESIA IN LOWER SEGMENT CAESAREAN SECTION. [cited 2021 Dec 18]; Available from: www.ijmedicines.com
- [Result] Ngan Kee WD, Lee SW, Ng FF, Tan PE, Khaw KS. Randomized double-blinded comparison of norepinephrine and phenylephrine for maintenance of blood pressure during spinal anesthesia for cesarean delivery. Anesthesiology. 2015 Apr;122(4):736-45. doi: 10.1097/ALN.0000000000000601. PMID 25635593
- [Result] Hasanin AM, Amin SM, Agiza NA, Elsayed MK, Refaat S, Hussein HA, Rouk TI, Alrahmany M, Elsayad ME, Elshafaei KA, Refaie A. Norepinephrine Infusion for Preventing Postspinal Anesthesia Hypotension during Cesarean Delivery: A Randomized Dose-finding Trial. Anesthesiology. 2019 Jan;130(1):55-62. doi: 10.1097/ALN.0000000000002483. PMID 30335625
- [Result] Wang X, Shen X, Liu S, Yang J, Xu S. The Efficacy and Safety of Norepinephrine and Its Feasibility as a Replacement for Phenylephrine to Manage Maternal Hypotension during Elective Cesarean Delivery under Spinal Anesthesia. Biomed Res Int. 2018 Dec 31;2018:1869189. doi: 10.1155/2018/1869189. eCollection 2018. PMID 30687737
- [Result] Xu C, Liu S, Qian D, Liu A, Liu C, Chen Y, Qi D. Preventive intramuscular phenylephrine in elective cesarean section under spinal anesthesia: A randomized controlled trial. Int J Surg. 2019 Feb;62:5-11. doi: 10.1016/j.ijsu.2018.12.014. Epub 2019 Jan 11. PMID 30639574
- [Result] Oh AY, Hwang JW, Song IA, Kim MH, Ryu JH, Park HP, Jeon YT, Do SH. Influence of the timing of administration of crystalloid on maternal hypotension during spinal anesthesia for cesarean delivery: preload versus coload. BMC Anesthesiol. 2014 May 16;14:36. doi: 10.1186/1471-2253-14-36. eCollection 2014. PMID 24920942
- [Result] Kinsella SM, Carvalho B, Dyer RA, Fernando R, McDonnell N, Mercier FJ, Palanisamy A, Sia ATH, Van de Velde M, Vercueil A; Consensus Statement Collaborators. International consensus statement on the management of hypotension with vasopressors during caesarean section under spinal anaesthesia. Anaesthesia. 2018 Jan;73(1):71-92. doi: 10.1111/anae.14080. Epub 2017 Nov 1. No abstract available. PMID 29090733
- [Result] Xu C, Liu S, Huang Y, Guo X, Xiao H, Qi D. Phenylephrine vs ephedrine in cesarean delivery under spinal anesthesia: A systematic literature review and meta-analysis. Int J Surg. 2018 Dec;60:48-59. doi: 10.1016/j.ijsu.2018.10.039. Epub 2018 Oct 31. PMID 30389535